CLINICAL TRIAL: NCT03079063
Title: Randomized, Multicenter, Single-dose, Cross-over, Double-blind Study Comparing the Pharmacokinetic of Biosimilar Eptacog Alfa With Novoseven®, in Patients With Congenital Factor VII Deficiency
Brief Title: Study Comparing the Pharmacokinetic of Biosimilar Eptacog Alfa With Novoseven®, in Patients With Congenital Factor VII Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AryoGen Pharmed Co. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: UGA2014-02
Record Dates: First submitted 2017-03-04; First posted 2017-03-14 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2020-07

CONDITIONS: Factor VII Deficiency
MeSH Terms: conditions — Factor VII Deficiency | interventions — recombinant FVIIa; Biosimilar Pharmaceuticals

STUDY DESIGN:
Intervention Model Description: Randomized, single dose, double blinded, two-way cross-over study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding is performed by an independent third party operator (nurse/pharmacist, unblinded), who will prepare undistinguishable syringes with patient's dosing and labeling. Central lab operators will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eptacog alfa biosimilar for PK (Experimental): Randomized, double-blind, single dose cross-over for PK, with 12 months follow up with eptacog alfa biosimilar provided for treatment of bleeding on demand - or - prophylaxis.
  Interventions: Biological: Eptacog alfa, biosimilar
- Novoseven (Active Comparator): Randomized, double-blind, single dose cross-over for PK, with 12 months follow up with eptacog alfa biosimilar provided for treatment of bleeding on demand - or - prophylaxis.
  Interventions: Biological: Novoseven

INTERVENTIONS:
Biological: Eptacog alfa, biosimilar — Either a single dose of eptacog alfa biosimilar 30 μg/kg and one single dose of NovoSeven 30 μg/kg, or vice versa, with doses separated by a washout period. Then, in an open follow up phase of 12 months, for every bleeding episode eptacog alfa biosimilar 30 μg/kg, on demand, for one of more days until resolution of bleeding, based on the Investigator's decision - or - prophylaxis with eptacog alfa biosimilar, with dose, frequency, and duration of treatment based on the Investigator's decision. The modality of treatment (on demand or prophylaxis) will be decided by the Investigator.
  Arms: Eptacog alfa biosimilar for PK
Biological: Novoseven — Either a single dose of eptacog alfa biosimilar 30 μg/kg and one single dose of NovoSeven 30 μg/kg, or vice versa, with doses separated by a washout period.
  Arms: Novoseven

SUMMARY:
The purpose of this multicentre, randomized, double blinded, single dose, two-way cross-over study, is to compare the pharmacokinetics (PK) of biosimilar eptacog alfa (activated) with Novoseven in 24 patients, adult and children (>12 years), not bleeding, with inherited coagulation factor VII (FVII) deficiency (FVII <1%). Patients will be randomized to receive either a single dose of eptacog alfa biosimilar 30 μg/kg and one single dose of NovoSeven 30 μg/kg, or vice versa, with doses separated by a washout period. All patients will be followed 12 months and will receive biosimilar eptacog alfa, on demand, for every bleeding episode that should occur - or - for prophylaxis, with the aim of monitoring of inhibiting antibody formation, lack of efficacy and collection of safety data.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of congenital, severe Factor VII deficiency (FVII <1%), with > 2 episodes of bleeding/year requiring treatment with FVII infusions, in non bleeding status.
* Patients for the Additional group for immunogenicity should be enrolled when in a bleeding episode requiring treatment with FVII.
* Male and female subjects
* Adult and children (>12 years)
* Written informed consent. For minor patients, parent/legal guardian will provide consent and, when possible, patient assent will also be obtained. For compromised patients their designated proxy must provide informed consent.

Exclusion Criteria:

* Any other type of congenital or acquired coagulopathy (except congenital Factor VII deficiency), such as: liver disease (hepatitis), vitamin k deficiency, uremia, malignancy.
* Antibodies against Factor VII
* Patients entering the PK Study Group who have not suspended prophylactic regimen with Novoseven or AryoSeven (biosimilar eptacog alfa) 3 days before starting the trial (receiving first dose of study medication).
* Patients entering the Additional Group for Immunogenicity study, only, who have been exposed to AryoSeven before starting study [patients who have received Novoseven (on demand or in prophylaxis) before starting study are allowed]
* Platelet count less than 100.000 platelets/μl (at screening visit)
* Patients who have received routine (prophylactic) treatment with rFVIIa in the period between screening visit (visit 1) and visit 2 of this study (first dose administration)
* Any clinical sign or known history of arterial thrombotic event or deep venous- thrombosis or pulmonary embolism
* HIV positive with current CD4+ count of less than 200/μl
* Liver Cirrhosis
* Known hypersensitivity to the study medication
* Parallel participation in another experimental drug trial.
* Parallel participation in another marketed drug trial that may affect the primary end point of the study.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Male and female
Enrollment: 24 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
Area under the plasma activity-time curve from time 0 to last quantifiable activity (AUClast) | Ten min before injection and 10 min, 20 min, 1h, 3h, 6h, 8h, 12h, 24h and 30h after injection, for both drug administered in the PK phase
  Measurement of plasma level of factor VII clotting activity (FVII:C) [one-stage clotting method using recombinant tissue factor preparation (STA-Deficient and STA-Neoplastin R; Diagnostica Stago, France)],
Maximum plasma concentration of the factor VII activity (Cmax). | Ten min before injection and 10 min, 20 min, 1h, 3h, 6h, 8h, 12h, 24h and 30h after injection, for both drug administered in the PK phase
  Measurement of plasma level of factor VII clotting activity (FVII:C) [one-stage clotting method using recombinant tissue factor preparation (STA-Deficient and STA-Neoplastin R; Diagnostica Stago, France)],

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time 0 to infinity (AUCinf) | Ten min before injection and 10 min, 20 min, 1h, 3h, 6h, 8h, 12h, 24h and 30h after injection, for both drug administered in the PK phase
  Measurement of plasma level of factor VII clotting activity (FVII:C) [one-stage clotting method using recombinant tissue factor preparation (STA-Deficient and STA-Neoplastin R; Diagnostica Stago, France)]
Time of Cmax (tmax) | Ten min before injection and 10 min, 20 min, 1h, 3h, 6h, 8h, 12h, 24h and 30h after injection, for both drug administered in the PK phase
  Measurement of plasma level of factor VII clotting activity (FVII:C) [one-stage clotting method using recombinant tissue factor preparation (STA-Deficient and STA-Neoplastin R; Diagnostica Stago, France)]
Fraction of the total AUCinf that was derived by extrapolation beyond tlast (AUCextra) | Ten min before injection and 10 min, 20 min, 1h, 3h, 6h, 8h, 12h, 24h and 30h after injection, for both drug administered in the PK phase
  Measurement of plasma level of factor VII clotting activity (FVII:C) [one-stage clotting method using recombinant tissue factor preparation (STA-Deficient and STA-Neoplastin R; Diagnostica Stago, France)]
First order rate constant associated with the terminal (log-linear) portion of the curve (λz) | Ten min before injection and 10 min, 20 min, 1h, 3h, 6h, 8h, 12h, 24h and 30h after injection, for both drug administered in the PK phase
  Measurement of plasma level of factor VII clotting activity (FVII:C) [one-stage clotting method using recombinant tissue factor preparation (STA-Deficient and STA-Neoplastin R; Diagnostica Stago, France)]
Elimination half-life (t½) | Ten min before injection and 10 min, 20 min, 1h, 3h, 6h, 8h, 12h, 24h and 30h after injection, for both drug administered in the PK phase
  Measurement of plasma level of factor VII clotting activity (FVII:C) [one-stage clotting method using recombinant tissue factor preparation (STA-Deficient and STA-Neoplastin R; Diagnostica Stago, France)]
Mean residence time (MRT) | Ten min before injection and 10 min, 20 min, 1h, 3h, 6h, 8h, 12h, 24h and 30h after injection, for both drug administered in the PK phase
  Measurement of plasma level of factor VII clotting activity (FVII:C) [one-stage clotting method using recombinant tissue factor preparation (STA-Deficient and STA-Neoplastin R; Diagnostica Stago, France)]
Clearance (CL) | Ten min before injection and 10 min, 20 min, 1h, 3h, 6h, 8h, 12h, 24h and 30h after injection, for both drug administered in the PK phase
  Measurement of plasma level of factor VII clotting activity (FVII:C) [one-stage clotting method using recombinant tissue factor preparation (STA-Deficient and STA-Neoplastin R; Diagnostica Stago, France)]
Volume of distribution (Vss) | Ten min before injection and 10 min, 20 min, 1h, 3h, 6h, 8h, 12h, 24h and 30h after injection, for both drug administered in the PK phase
  Measurement of plasma level of factor VII clotting activity (FVII:C) [one-stage clotting method using recombinant tissue factor preparation (STA-Deficient and STA-Neoplastin R; Diagnostica Stago, France)]
Clinical response in controlling acute bleeding. | 2, 6 and 12 hours post infusion (last dose of Eptacog alfa Biosimilar)
  Rated by the treating physician using a 4 point scale (Excellent, Good, Moderate, None).
Immunogenicity | On plasma samples obtained at screening visit, before the second dose/second drug administration, and then every 3 months for a year.
  The modified Nijmegen method of the Bethesda assay
Adverse Events | Adverse events (AEs) will be monitored throughout the trial, from the first dose administered up to 12 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Iacobelli, MD, Study Director
Locations (2):
- Iran (2):
  - Hemophilia Center - Hematology & Oncology Dept. Shiraz University of Medical Science, Shiraz
  - Comprehensive Hemophilia Care Center, Tehran

IPD SHARING:
Plan to Share IPD: Undecided